CLINICAL TRIAL: NCT02104245
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Pulmaquin® in the Management of Chronic Lung Infections With Pseudomonas Aeruginosa in Patients With Non-Cystic Fibrosis Bronchiectasis, Including 28 Day Open-Label Extension
Brief Title: Phase 3 Study With Ciprofloxacin Dispersion for Inhalation in Non-CF Bronchiectasis (ORBIT-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aradigm Corporation (Industry)
Collaborators: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Organization: Savara Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARD-3150-1202
Record Dates: First submitted 2014-03-28; First posted 2014-04-04 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Non Cystic Fibrosis Bronchiectasis
Keywords: Non Cystic Fibrosis Bronchiectasis, Pulmaquin, Ciprofloxacin, Pseudomonas aeruginosa
MeSH Terms: conditions — Pseudomonas Infections | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciprofloxacin dispersion for inhalation (Experimental): Liquid mixture of liposomally encapsulated and unencapsulated ciprofloxacin
  Interventions: Drug: Ciprofloxacin dispersion for inhalation
- Placebo (Placebo Comparator): Liquid formulation of empty liposomes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin dispersion for inhalation
  Arms: Ciprofloxacin dispersion for inhalation
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study (ARD-3150-1202, ORBIT-4) will evaluate the safety and efficacy of inhaled Pulmaquin (ciprofloxacin dispersion for inhalation) compared to inhaled placebo in subjects who have a confirmed diagnosis of non-cystic fibrosis (non-CF) bronchiectasis with a history of pulmonary exacerbations and chronic P. aeruginosa infections.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of non-CF bronchiectasis
* History of P. aeruginosa respiratory infections
* At least two pulmonary exacerbations treated with antibiotics in the previous year

Exclusion Criteria:

* Have a clinical diagnosis of CF
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Time to first pulmonary exacerbation (from baseline) | 48 weeks

CONTACTS AND LOCATIONS:
Locations (95):
- United States (25):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sacramento, California
  - San Diego, California
  - Torrance, California
  - Danbury, Connecticut
  - Miami, Florida
  - Orlando, Florida
  - Winter Park, Florida
  - Decatur, Georgia
  - Duluth, Georgia
  - Port Huron, Michigan
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Summit, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Chapel Hill, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Rock Hill, South Carolina
  - Spartanburg, South Carolina
  - Tyler, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (4):
  - Greenslopes, Queensland
  - Adelaide, South Australia
  - Nedlands, Western Australia
  - Perth, Western Australia
- Canada (4):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Windsor, Ontario
  - Saint-Jérôme, Quebec
- France (6):
  - Créteil
  - Grenoble
  - Nice
  - Pessac
  - Rouen
  - Toulouse
- Georgia (2):
  - Kutaisi
  - Tbilisi
- Hungary (4):
  - Budapest
  - Nyíregyháza
  - Székesfehérvár
  - Törökbálint
- Israel (4):
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (7):
  - Avellino
  - Napoli
  - Parma
  - Pisa
  - San Gerardo
  - Terni
  - Trieste
- New Zealand (3):
  - Otahuhu, Auckland
  - Hamilton, Waikato Region
  - Tauranga
- Peru (4):
  - Jesus Maria, Lima region
  - La Victoria, Lima region
  - Pueblo Libre, Lima region
  - San Juan de Miraflores, Lima region
- Poland (4):
  - Bialystok
  - Krakow
  - Ruda Śląska
  - Warsaw
- Romania (5):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
- Serbia and Montenegro (4):
  - Belgrade
  - Knez Selo
  - Kragujevac
  - Sremska Kamenica
- South Korea (3):
  - Suwon, Gyeonggi-do
  - Daegu
  - Seoul
- Spain (4):
  - A Coruña
  - Barcelona
  - Lleida
  - Valencia
- United Kingdom (12):
  - Stockton-on-Trees, Cleveland
  - Wigan, Greater Manchester
  - Cambridge
  - Colchester
  - Cottingham
  - Lancaster
  - Leeds
  - London
  - Manchester
  - North Sheilds
  - Southampton
  - Telford

REFERENCES:
- [Derived] Chalmers JD, Cipolla D, Thompson B, Davis AM, O'Donnell A, Tino G, Gonda I, Haworth C, Froehlich J. Changes in respiratory symptoms during 48-week treatment with ARD-3150 (inhaled liposomal ciprofloxacin) in bronchiectasis: results from the ORBIT-3 and -4 studies. Eur Respir J. 2020 Oct 22;56(4):2000110. doi: 10.1183/13993003.00110-2020. Print 2020 Oct. PMID 32554534
- [Derived] Haworth CS, Bilton D, Chalmers JD, Davis AM, Froehlich J, Gonda I, Thompson B, Wanner A, O'Donnell AE. Inhaled liposomal ciprofloxacin in patients with non-cystic fibrosis bronchiectasis and chronic lung infection with Pseudomonas aeruginosa (ORBIT-3 and ORBIT-4): two phase 3, randomised controlled trials. Lancet Respir Med. 2019 Mar;7(3):213-226. doi: 10.1016/S2213-2600(18)30427-2. Epub 2019 Jan 15. PMID 30658914